CLINICAL TRIAL: NCT01341808
Title: Immunogenicity of Hepatitis A Vaccine in Patients With Inflammatory Bowel Disease
Brief Title: Immunogenicity of Hepatitis A Vaccine in Inflammatory Bowel Disease (IBD) Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Suk-Kyun Yang, Professor, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2011-0047
Record Dates: First submitted 2011-04-25; First posted 2011-04-26 (Estimated); Last update posted 2013-03-19 (Estimated); Status verified 2013-03

CONDITIONS: Inflammatory Bowel Disease; Crohn's Disease; Ulcerative Colitis; Hepatitis A
Keywords: Crohn's disease; Ulcerative colitis; Hepatitis A; vaccine
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative; Hepatitis A | interventions — epaxal berna

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IBD patients (Experimental): Patients diagnosed with IBD
  -> receive Epaxal Berna (virosomal hepatitis A vaccine)
  Interventions: Biological: Epaxal Berna (virosomal hepatitis A vaccine)

INTERVENTIONS:
Biological: Epaxal Berna (virosomal hepatitis A vaccine) — standard 0.5 mL dose of Epaxal Berna (virosomal hepatitis A vaccine) given at Day 0, Month 6.
  Other Names: Epaxal Berna

SUMMARY:
The purpose of this study is to measure the immune response in 18-40 year old IBD patients after receiving the hepatitis A vaccine.

DETAILED DESCRIPTION:
The spread of hepatitis A has prompted the need for vaccination against this virus. It is uncertain that IBD patients can achieve a truly protective response after vaccination. The efficacy and safety of hepatitis A vaccination have not been evaluated in this population of patients. We would like to estimate the efficacy and safety of vaccination against hepatitis A in patients with IBD.

ELIGIBILITY:
Inclusion Criteria:

1. Patients suffering from inflammatory bowel disease: Crohn's disease/Ulcerative colitis
2. Age 18-40
3. Willing to provide informed consent

Exclusion Criteria:

1. Have history of vaccination to hepatitis A
2. Have other autoimmune disease
3. Have any malignancy
4. Have acute infectious disease
5. Unwilling to provide consent

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 493 (Actual)
Dates: Start 2011-04; Primary Completion 2013-02 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
antibody titer to hepatitis A vaccine | Month 7

SECONDARY OUTCOMES:
vaccine-associated adverse events and side effects | within the first 30 days after first vaccination
vaccine-associated adverse events and side effects | within the first 30 days after second vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Suk-Kyun Yang, M.D., Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

REFERENCES:
- [Background] D'Acremont V, Herzog C, Genton B. Immunogenicity and safety of a virosomal hepatitis A vaccine (Epaxal) in the elderly. J Travel Med. 2006 Mar-Apr;13(2):78-83. doi: 10.1111/j.1708-8305.2006.00001.x. PMID 16553593
- [Background] Hou JK, Velayos F, Terrault N, Mahadevan U. Viral hepatitis and inflammatory bowel disease. Inflamm Bowel Dis. 2010 Jun;16(6):925-32. doi: 10.1002/ibd.21284. PMID 20480515
- [Derived] Park SH, Yang SK, Park SK, Kim JW, Yang DH, Jung KW, Kim KJ, Ye BD, Byeon JS, Myung SJ, Kim JH. Efficacy of hepatitis A vaccination and factors impacting on seroconversion in patients with inflammatory bowel disease. Inflamm Bowel Dis. 2014 Jan;20(1):69-74. doi: 10.1097/01.MIB.0000437736.91712.a1. PMID 24284413